CLINICAL TRIAL: NCT06250218
Title: Does the Intervention Video Interactive Guidance (VIG) Have an Impact on the Development of the Language and Sociocognitive Skills of Children Aged Between 2 and 5 With Identified Language Delays?
Brief Title: Using Video Interaction Guidance (VIG) With Children Who Have Language Delays.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sheffield (Other)
Responsible Party: Principal Investigator, Emma J Harvey, Educational Visitor (Dumfries and Galloway Council). Student (University of Sheffield)., University of Sheffield
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 001
Record Dates: First submitted 2024-01-18; First posted 2024-02-09 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Language Development Disorders
MeSH Terms: conditions — Language Development Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Group (Experimental): The group will receive the intervention Video Interaction Guidance.
  Interventions: Other: Video Interactive Guidance (VIG)

INTERVENTIONS:
Other: Video Interactive Guidance (VIG) — Video interaction guidance (VIG) is a video feedback intervention through which a "guider" helps a client to enhance communication within relationships. The client is guided to analyse and reflect on video clips of their own interactions.

SUMMARY:
The study aims to explore whether the intervention Video Interactive Guidance (VIG) has an impact on the development of the language and sociocognitive skills of children aged between 2 and 5 with identified language delays. The study is expected to take the form of a small mixed methods case study of AB design and is anticipated to involve 4 participants.

DETAILED DESCRIPTION:
The study will take the form of a small mixed methods case study of AB design and is expected to involve 4 participants. These participants are children aged between 2 and 4 who have all been referred to the Educational Visiting Service, a specialist branch of Early Years Education in Dumfries and Galloway local authority, within which the researcher currently works as an Educational Visitor. The children's key workers at nursery will be involved in the delivery of this video-based intervention and it is from both the child's parents/carers and them that informed consent to participate will be sought. Any identifying text based personal information and gathered assessment data will be coded to preserve the anonymity of the participants. Consent to store and share original, unaltered audio-visual recordings with research supervisors will be gained from the participant's parents and key workers. These recordings will be thematically analysed and coded before they are included in the final project, again to preserve the anonymity of the participants. Any original recordings made will be securely stored on the researcher's university managed Google Drive until the project is complete and then deleted. As the researcher is currently working towards full accreditation from aVIGUK, they have been appointed an aVIGUK accredited supervisor for the duration of this project. Alongside the University research supervisors, they will be responsible for overseeing the project and will carry out regular supervision meetings with the researcher. This will involve the reviewing of the researchers filmed intervention sessions to ensure that the researcher adheres to the aVIGUK approved method of delivering the intervention, as well as corroborating and cross-checking the researcher's collected data.

Each of the participants will receive the intervention Video Interaction Guidance (VIG) with their key worker at nursery. Three norm-referenced standardised tests will be carried out at T1 (pre-intervention stage, 6 weeks before the intervention takes place), T2 (immediately prior to the intervention taking place) and T3 (immediately after the intervention takes place). The tests that will be carried out are the Renfrewshire Action Picture test (measuring expressive language, specifically information and grammar), the Renfrewshire Expressive Vocabulary test (measuring expressive vocabulary, specifically the extent to which objects can be named verbally from their picture) and the Hogrefe Early Sociocognitive Battery (measuring early sociocognitive skills, (specifically their social responsiveness, joint attention and symbolic comprehension). These assessments will be scored by the researcher but will also be filmed to allow for an independent evaluation to be carried out by an aVIGUK appointed supervisor. This will be done by sampling the videos at random, a second scoring being carried out by the aVIG UK approved supervisor and the scores compared. The purpose of this is to limit the impact of researcher bias and improve the internal validity of the study. MORS (see Appendix A) and Belfast (see Appendix B) assessments will also be carried out for each of the children at T1, T2 and T3. These assessments are not standardised but will provide data similar in style to the qualitative data provided by semi-structured interviews and will be analysed thematically. The final method of data collection will be an analysis of the first and final sessions of each of the participants. These will be coded in the same way as the Early Sociocognitive Battery with an emphasis on social responsiveness, joint attention and symbolic comprehension. As previously, samples of this analysis will be cross-evaluated by an aVIGUK appointed supervisor to improve the internal validity of the study.

ELIGIBILITY:
Inclusion Criteria:

* Identified language delay (identified by participants Health Visitor through ASQ-3 assessment.

Exclusion Criteria:

* No identified language delay

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 4 (Estimated)
Dates: Start 2024-02 (Estimated); Primary Completion 2024-08 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Social Responsiveness | 5 weeks
  A subtest of the Early Sociocognitive Battery Assessment will be used to determine whether there was a change in the participant's social responsiveness after the intervention.
Joint Attention | 5 weeks
  A subtest of the Early Sociocognitive Battery Assessment will be used to determine whether there was a change in the participant's joint attention after the intervention.
Symbolic Comprehension | 5 weeks
  A subtest of the Early Sociocognitive Battery Assessment will be used to determine whether there was a change in the participant's symbolic comprehension after the intervention.
Expressive Language - Information | 5 weeks
  A subtest of the Renfrew Action Picture Test will be used to determine whether there was a change in the participant's expressive language (information) after the intervention.
Expressive Language - Grammar | 5 weeks
  A subtest of the Renfrew Action Picture Test will be used to determine whether there was a change in the participant's expressive language (grammar) after the intervention.
Expressive Vocabulary | 5 weeks
  A subtest of the Renfrewshire Expressive Vocabulary Test will be used to determine whether there was a change in the participant's expressive vocabulary after the intervention.

IPD SHARING:
Plan to Share IPD: No
Any identifying text based personal information and gathered assessment data will be coded to preserve the anonymity of the participants. Consent to store and share original, unaltered audio-visual recordings with research supervisors will be gained from the participant's parents and key workers. These recordings will be thematically analysed and coded before they are included in the final project, again to preserve the anonymity of the participants.